CLINICAL TRIAL: NCT00206999
Title: Early Information Processing in Healthy Controls: Studies on the Relation Between Two Different Paradigms (PPI and P50ERP) and Effects of Pharmacological Interventions
Brief Title: The Effect of Imipramine on Early Information Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birte Glenthoj (Other)
Collaborators: University of Copenhagen (Other); Glostrup University Hospital, Copenhagen (Other); The Danish Medical Research Council (Other); Lundbeck Foundation (Other)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 363052-2; KF 01-305/99; KF 11-061/03; KF 11-068/03; KF 11-096/04
Record Dates: First submitted 2005-09-11; First posted 2005-09-21 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Volunteers
Keywords: Psychophysiology; PPI; P50 suppression; Imipramine
MeSH Terms: interventions — Imipramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: imipramine

INTERVENTIONS:
Drug: imipramine — Either 50 mg of imipramine or placebo will be administered to healthy male volunteers

SUMMARY:
We wanted to compare the relation of two different psychophysiological paradigms (PrePulse Inhibition of the startle response = PPI and P50 suppression) to each other. Additionally, we wanted to test the effect of the combined serotonin- and noradrenaline re-uptake inhibitor, imipramine, on these measures. The primary hypothesis was that PPI and P50 gating would not correlate with each other at baseline. The secondary hypothesis was that increased noradrenergic and serotonergic activity would disrupt PPI as well as P50 gating.

DETAILED DESCRIPTION:
Schizophrenic patients exhibit impairments in filtering of sensory information, as can be assessed by use of prepulse inhibition (PPI) of the acoustic startle response and P50 suppression paradigms. In the treatment of negative symptoms or depressive syndromes during the course of schizophrenia antidepressants are often combined with antipsychotic medication. However, antidepressants increase monoaminergic activity, of which in turn it has been suggested to decrease sensory gating, although these presumptions are mostly based on results from animal studies. Currently, little is known about monoaminergic modulation of sensory filtering in humans, and the few reports that can be found in literature show discrepancies with animal studies. The current study was designed to study the effects of increased monoaminergic activity on sensory filtering and habituation of healthy volunteers. In a double-blind, placebo controlled cross-over design, twenty healthy male volunteers will receive either placebo or a dose of 50 mg of imipramine (a dual acting antidepressant), after which they will be tested in a P50 suppression-, a PPI-, and a habituation of the startle reflex paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Good Physical and Mental Health meeting criteria "never mentally ill", which will be evaluated with a medical history checklist, ECG
* Non smokers

Exclusion Criteria:

* Current use of any medication
* Any subject who has received any investigational medication within 30 days prior to the start of this study
* History of neurologic illness
* History of psychiatric illness in first-degree relatives, evaluated with DSM-IV criteria
* History of alcohol and drug abuse. Positive urine screening for amphetamine, cocaine, cannabis, or ecstasy.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Sensory gating | Once, 1 hour after administration of capsule

SECONDARY OUTCOMES:
PPI of the startle reflex | once, one hour after administration
P50 suppression | once, one hour after administration

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthoj, MD, DMSc., Study Director — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychaitric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- See also: Center for Neuropsychiatric Schizophrenia Research (CNSR) — http://www.cnsr.dk